CLINICAL TRIAL: NCT03959514
Title: Phase I Single Dose, Randomised, Double-blind, Three-way Cross Over, Glucose Clamp Study Investigating the PK/PD and Safety of Arecor Ultra-rapid Insulin Aspart (AT247) in Comparison to NovoRapid® and Fiasp® in Participants With Type I Diabetes Mellitus (T1DM).
Brief Title: AT247, NovoRapid® and Fiasp® in Glucose Clamp Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arecor Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARE-247-101
Record Dates: First submitted 2019-05-13; First posted 2019-05-22 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AT247 (Experimental): Single subcutaneous injection 0.3 U/Kg
  Interventions: Biological: NovoRapid; Biological: Fiasp; Biological: AT247
- NovoRapid (Active Comparator): Single subcutaneous injection 0.3 U/Kg
  Interventions: Biological: NovoRapid; Biological: Fiasp; Biological: AT247
- Fiasp (Active Comparator): Single subcutaneous injection 0.3 U/Kg
  Interventions: Biological: NovoRapid; Biological: Fiasp; Biological: AT247

INTERVENTIONS:
Biological: NovoRapid — Rapid acting prandial insulin aspart
  Other Names: NovoLog
Biological: Fiasp — Fast acting prandial insulin aspart
Biological: AT247 — Ultra rapid acting prandial insulin aspart

SUMMARY:
A Phase I, randomised, single-centre, double-blind, single-dose, three period, balanced cross over study in a glucose clamp setting. The study compares the pharmacodynamic, pharmacokinetic and safety characteristics of AT247, NovoRapid® and Fiasp® in male participants with type I diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria include:

1. Diagnosis type I Diabetes Mellitus for at least 12 months
2. Receiving treatment with multiple daily insulin injections or insulin pump therapy for at least 12 months
3. Fasting C-peptide concentration ≤8.5% (≤69 mmol/mol) at screening
4. BMI 18.5-35.0 kg/m2

Exclusion Criteria include:

1. known or suspected hypersensitivity to Investigational Medicinal Products
2. clinically significant concomitant disease or abnormal lab values
3. supine systolic BP outside range 95-140 mmHg and/or diastolic BP greater than 90 mmHg

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate-time curve of insulin aspart | 0-60 minutes

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve from 0-60 minutes | 0-60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Graz, Austria

REFERENCES:
- [Derived] Svehlikova E, Mursic I, Augustin T, Magnes C, Gerring D, Jezek J, Schwarzenbacher D, Ratzer M, Wolf M, Howell S, Zakrzewski L, Urschitz M, Tschapeller B, Gatschelhofer C, Feichtner F, Lawrence F, Pieber TR. Pharmacokinetics and Pharmacodynamics of Three Different Formulations of Insulin Aspart: A Randomized, Double-Blind, Crossover Study in Men With Type 1 Diabetes. Diabetes Care. 2021 Feb;44(2):448-455. doi: 10.2337/dc20-1017. Epub 2020 Dec 16. PMID 33328285